CLINICAL TRIAL: NCT05575973
Title: A Prospective, Single-arm, Multicenter Clinical Study of Mitoxantrone Hydrochloride Liposome Combined With Rituximab and Lenalidomide in the Treatment of Relapsed and Refractory Diffuse Large B-cell Lymphoma
Brief Title: Mitoxantrone Hydrochloride Liposome Combined With Rituximab and Lenalidomide (M+R2) in Patients With Relapsed and Refractory Diffuse Large B-Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jianfeng Zhou (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Jianfeng Zhou, Director, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DED-DLBCL-K03
Record Dates: First submitted 2022-09-28; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- mitoxantrone hydrochloride liposome (Experimental): Patients with relapsed and refractory diffuse large B-cell lymphoma (DLBCL) will receive sequentially mitoxantrone hydrochloride liposome in combination with rituximab and lenalidomide for up to 6 cycles (28 days per cycle).
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome; Drug: Rituximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome — Drug: Mitoxantrone hydrochloride liposome (20 mg/m2) will be administered by an intravenous infusion on day 1 of each 28-day cycle.
Drug: Rituximab — Drug: Rituximab (375 mg/m2) will be administered by an intravenous infusion on day 1 of each 28-day cycle.
Drug: Lenalidomide — Drug: Lenalidomide (25 mg) will be taken orally from day 1 to day 8 of each 28-day cycle.

SUMMARY:
To evaluate the safety and efficacy of mitoxantrone hydrochloride liposome in combination with rituximab and lenalidomide in the treatment of relapsed and refractory diffuse large B-cell lymphoma (DLBCL).

DETAILED DESCRIPTION:
This is a prospective, single-arm, multicenter phase Ⅱ clinical study to evaluate the safety and efficacy of mitoxantrone hydrochloride liposome in combination with rituximab and lenalidomide in patients with relapsed and refractory diffuse large B-cell lymphoma (DLBCL). Mitoxantrone hydrochloride liposome will be given on day 1 at the dose of 20 mg/m2 and be combined with rituximab and lenalidomide. A maximum of 6 cycles of therapy are planned.

ELIGIBILITY:
Inclusion Criteria:

* 1.Subjects fully understand and voluntarily participate in this study and sign the informed consent form (ICF);
* 2.60-75 years old;
* 3.Expected survival ≥ 3 months;
* 4.Subjects with histologically confirmed diagnosis of relapsed and refractory diffuse large B-cell lymphoma who have received at least 4 cycles of first-line chemotherapy including rituximab and anthracyclines; Relapsed lymphoma is defined as the lymphoma that relapse after obtaining complete response (CR) after initial chemotherapy; Refractory lymphoma subjects meet one of the following conditions: 1) The tumor shrinks <50% or disease progression after 4 cycles of standard chemotherapy,; 2) CR after standard chemotherapy, but relapse within half a year; 3) 2 or more relapses after CR; 4) relapse after hematopoietic stem cell transplantation;
* 5.Subjects who are not eligible for transplantation or do not plan to undergo transplantation at the beginning of the study;
* 6.ECOG Performance Status: 0-2;
* 7.Subjects must have at least one evaluable or measurable lesion per lugano2014 criteria: for lymph node lesions, the length should be > 1.5cm; For non-lymph node lesions, the length should be > 1.0cm;
* 8.Bone marrow function: Absolute neutrophil count ≥1.5×109/L, Platelet count ≥75×109/L, Hemoglobin ≥ 80g/L (Absolute neutrophil can be relaxed to ≥ 1.0×109/L, Platelet count can be relaxed to ≥50×109/L, Hemoglobin can be relaxed to ≥75 g/L in subjects with poor bone-marrow reserve);
* 9.Liver and kidney function: serum creatinine ≤ 1.5×ULN (upper limit of normal); AST and ALT ≤ 2.5×ULN (≤ 5×ULN for subjects with liver metastases); total bilirubin ≤ 1.5×ULN (≤ 3×ULN for subjects with liver metastases).

Exclusion Criteria:

* 1. The subject had previously received any of the following anti-tumor treatments:

  1. Subjects who have been treated with mitoxantrone or mitoxantrone liposomes;
  2. Previously received doxorubicin or other anthracycline treatment, and the total cumulative dose of doxorubicin was more than 360 mg/m2 (1 mg doxorubicin equivalent to 2 mg epirubicin);
  3. Subjects who received anti-tumor treatment (including chemotherapy, targeted therapy, glucocorticoid, traditional Chinese medicine with anti-tumor activity, etc.) or participated in other clinical trials and received trial drugs within 4 weeks or 5 T1/2s before the first administration of the study drugs;
  4. Subjects who received lenalidomide.
* 2.Subjects with refractory lymphoma meet one of the following criteria: 1) Tumors assessed as SD/PD after ≥2 lines of chemotherapy; 2) Subjects relapse within 6 months after transplantation.
* 3.Hypersensitivity to any study drug or its components;
* 4.Uncontrolled systemic diseases (such as active infection, uncontrolled hypertension, diabetes, etc.)
* 5.Heart function and disease meet one of the following conditions:

  1. Long QTc syndrome or QTc interval > 480 ms;
  2. Complete left bundle branch block, grade II or III atrioventricular block;
  3. Serious and uncontrolled arrhythmias requiring drug treatment;
  4. New York Heart Association grade ≥ III;
  5. Cardiac ejection fraction (LVEF)< 50%;
  6. A history of myocardial infarction, unstable angina pectoris, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, a history of clinically serious pericardial disease, or ECG evidence of acute ischemia or active conduction system abnormalities within 6 months before recruitment.
* 6.Hepatitis B and hepatitis C active infection (plus HBV DNA if one positive for hepatitis B surface antigen or core antibody and HBV DNA more than 1×103 copy/mL excluded; plus HCV RNA if hepatitis C antibody positive and HCV RNA more than 1×103 copy/mL exclude)
* 7.Baseline B-type pro-brain natriuretic peptide (NT-proBNP) > 1800pg/ml, troponin I (cTnI) > ULN of our center, and the retest data is still higher than the above range after three days;
* 8.Human immunodeficiency virus (HIV) infection (HIV antibody positive);
* 9.Subjects with other malignant tumors past or present (except for non-melanoma skin basal cell carcinoma, breast/cervical carcinoma in control, and other malignant tumors that have been effectively controlled without treatment within the past five years);
* 10.Subjects suffering from primary or secondary central nervous system (CNS) lymphoma or a history of CNS lymphoma at the time of recruitment;
* 11.Unsuitable subjects for this study determined by the investigator.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-10-10 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | through study completion, an average of 2 year
  To investigate the preliminary antitumor efficacy

SECONDARY OUTCOMES:
Progression free survival (PFS) | through study completion, an average of 2 year
  To investigate the preliminary antitumor efficacy
Duration of relief (DOR) | through study completion, an average of 2 year
  To investigate the preliminary antitumor efficacy
Disease Control Rate (DCR) | through study completion, an average of 2 year
  To investigate the preliminary antitumor efficacy
Best of response (BOR) | 6-8 weeks
  To investigate the preliminary antitumor efficacy
Safety endpoint: The incidence and severity of AE and SAE Safety endpoint: The incidence and severity of AE and SAE Safety endpoint:The incidence and severity of AE and SAE | through study completion, an average of 2 year
  To identify the incidence and severity of AE and SAE (NCI CTCAE v5.0)

OTHER OUTCOMES:
Efficacy assessed by IgNGS | through study completion, an average of 2 year
  Efficacy assessed by IgNGS
Other metrics that researchers are interested | through study completion, an average of 2 year
  Other metrics that researchers are interested

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China